CLINICAL TRIAL: NCT02087371
Title: Prognosis Factors of Cardiac Complications After Liver Transplantation
Acronym: PROCOM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOR12132
Record Dates: First submitted 2014-01-22; First posted 2014-03-14 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Hepatopathy
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and urines samples will be collected on 3 separate days (inclusion in the study, the day before liver transplantion and 7 days after).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Included patients: Patients with end-stage liver failure and registered on transplantation list.

SUMMARY:
This is a prospective, multicenter, non-interventional, observational study of a cohort with a biological plasma and urine samples collection for the study of prognosis factors of cardiac complications after liver transplantation

DETAILED DESCRIPTION:
Liver transplantation (LT) is the standard treatment for chronic or acute hepatic insufficiency with 87% of one-year survival. Cardiovascular complications are common after LT with an incidence at 6 months ranging between 25 and 50 %. These complications are associated with significant morbidity and represents the third cause of post LT mortality. Myocardial perfusion imaging or stress echocardiography, used for preoperative cardiovascular evaluation, are not enough efficient to predict the risk of post LT cardiovascular complications. However, to improve the prediction capacity of cardiovascular disease is fundamental in order to better select the candidates for LT or to develop preventive strategies. Such a strategy could reduce the morbidity and mortality from cardiovascular diseases after LT and improve the results of LT. Cardiovascular biomarkers such as troponin or natriuretic peptide are known to be predictive factors of postoperative cardiovascular complications in non cardiac surgery. The use of biomarkers in combination with conventional tests could improve the preoperative prediction of post LT cardiovascular complications.

Hypothesis: The preoperative biomarkers dosage could improve the prediction of cardiovascular complications occurring in the year after LT.

ELIGIBILITY:
Inclusion criteria:

- Patients older than 18 years, on list for LT because of chronic hepatic disease.

Non-inclusion criteria:

- emergency LT, patient under guardianship or trusteeship.

Secondary exclusion criteria:

* Patient out of list before liver transplant because of his death, his improvement, the existence of a contraindication
* Patient not presenting laboratory tests older than 1 year at the liver transplantaion.
* Patient included for over 2 years at the time of Liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage liver failure and registered on transplantation list can participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Cardiovascular complications | 1 year after liver transplantation
  Identify risk factors for occurrence of cardiovascular complications in the year following the transplantation.
  Cardiovascular complications include myocardial infarction, increase of cardiac troponin, cardiogenic pulmonary edema, cardiogenic shock, ventricular or supraventricular arrhythmia requiring treatment, de novo arterial hypertension and death of cardiac cause.

SECONDARY OUTCOMES:
Describe prospectively cardiovascular complications after liver transplantation | 1 year after liver transplantation
Assess the impact of these complications on morbidity and mortality in intensive care at J28 and 1 year. | 1 year after liver transplantation
Gather a biological plasma and urine samples collection for study of new biomarkers. | 7 days after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Catherine PAUGAM BURTZ, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France

IPD SHARING:
Plan to Share IPD: No